CLINICAL TRIAL: NCT05394142
Title: A Phase II, Randomised, Multi-centric, Multi-national Clinical Trial to Evaluate the Efficacy, Tolerability, and Safety of a Fixed Dose Combination of Spironolactone, Pioglitazone & Metformin (SPIOMET) for Adolescent Girls and Young Adult Women (AYAs) With Polycystic Ovary Syndrome (PCOS)
Brief Title: A Clinical Trial to Evaluate the Efficacy, Tolerability, and Safety of a Fixed Dose Combination of Spironolactone, Pioglitazone & Metformin (SPIOMET) in Polycystic Ovary Syndrome (PCOS)
Acronym: SPIOMET4HEALTH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPIOMET4HEALTH; 2021-003177-58 (EudraCT Number)
Record Dates: First submitted 2022-05-09; First posted 2022-05-27 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: polycystic ovary syndrome; spironolactone; pioglitazone; metformin; peadiatric; PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Pioglitazone; Spironolactone; Metformin

STUDY DESIGN:
Intervention Model Description: This is a multi-centre, multi-national, double-blinded, placebo-controlled, parallel, randomised Phase 2 clinical trial with four subgroups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 - Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Arm 1 - PIO (Experimental): Pioglitazone
  Interventions: Drug: Pioglitazone
- Arm 1 - SPIO (Experimental): Spironolactone and Pioglitazone
  Interventions: Drug: Pioglitazone; Drug: Spironolactone
- Arm 1 - SPIOMET (Experimental): Spironolactone, Pioglitazone and Metformin
  Interventions: Drug: Pioglitazone; Drug: Spironolactone; Drug: Metformin

INTERVENTIONS:
Drug: Placebo — Comparator arm with placebo
  Arms: Arm 1 - Placebo
Drug: Pioglitazone — Pioglitazone 7.5 mg/day
  Other Names: PIO
  Arms: Arm 1 - PIO; Arm 1 - SPIO; Arm 1 - SPIOMET
Drug: Spironolactone — Spironolactone 50 mg/day
  Other Names: S
  Arms: Arm 1 - SPIO; Arm 1 - SPIOMET
Drug: Metformin — Metformin 850 mg/day
  Other Names: MET
  Arms: Arm 1 - SPIOMET

SUMMARY:
This is a multi-centre, multi-national, double-blinded, placebo-controlled, parallel, randomised Phase II clinical trial to evaluate the efficacy, tolerability, and safety of a fixed dose combination of Spironolactone, Pioglitazone and Metformin (SPIOMET) for adolescent girls and young adult women with polycystic ovary syndrome.

Study description: Currently, there is no European Medicines Agency /U.S. Food and Drug Administration (FDA)-approved therapy for polycystic ovary syndrome in adolescent girls and young adult women. Oral contraceptives (OCs) are prescribed off-label to approximately 98% of AYAs with PCOS, including those without pregnancy risk. OCs alleviate key symptoms by inducing a pharmacological combination of anovulatory subfertility, regular pseudo-menses, and extreme elevations of sex hormone-binding globulin (SHBG), but OCs do not revert the underlying pathophysiology, and patients remain at risk for post-treatment subfertility and possibly, for lifelong co-morbidities.

Given the key role of hepato-visceral fat excess in the pathogenesis of PCOS, the prime aim of the treatment should be to achieve a preferential loss of central fat, which should in turn normalise the entire PCOS phenotype. Recent evidence disclosed that a treatment consisting of a fixed low-dose combination of two insulin sensitisers [pioglitazone (PIO) and metformin (MET), with different modes of action], and one mixed anti-androgen and anti-mineralocorticoid (spironolactone), was superior to an OC in normalising the PCOS phenotype, including ovulation rates and hepato-visceral fat.

The study's main goals are to assess the efficacy, tolerability and safety of a new treatment (SPIOMET) for adolescent girls and young adult women with polycistic ovarian syndrome; the comparison (in this order) of each SPIOMET, spironolactone and pioglitazone (SPIO) and PIO over placebo; and in addition, the comparison of SPIOMET over PIO and over SPIO (in this order).

Primary Objective: To test the efficacy of SPIOMET in normalising ovulation rate in adolescents and young adult women with PCOS.

Secondary Objectives: To test the efficacy of SPIOMET in normalising the endocrine-metabolic status, to describe the drug safety profile and to assess the adherence and subjective acceptability, as well as the quality of life of the participating subjects.

DETAILED DESCRIPTION:
This is a multi-centre, multi-national, double-blinded, placebo-controlled, parallel, randomised Phase II clinical trial to evaluate the efficacy, tolerability, and safety of a fixed dose combination of Spironolactone, Pioglitazone and Metformin (SPIOMET) for adolescent girls and young adult women (AYAs) with polycystic ovary syndrome (PCOS).

Study description: Currently, there is no European Medicines Agency (EMA)/U.S. Food and Drug Administration (FDA)-approved therapy for PCOS in AYAs. Oral contraceptives (OCs) are prescribed off-label to approximately 98% of AYAs with PCOS, including those without pregnancy risk. OCs alleviate key symptoms by inducing a pharmacological combination of anovulatory subfertility, regular pseudo-menses, and extreme elevations of sex hormone-binding globulin (SHBG), but OCs do not revert the underlying pathophysiology, and patients remain at risk for post-treatment subfertility and possibly, for lifelong co-morbidities.

Given the key role of hepato-visceral fat excess in the pathogenesis of PCOS, the prime aim of the treatment should be to achieve a preferential loss of central fat, which should in turn normalise the entire PCOS phenotype. Recent evidence disclosed that a treatment consisting of a fixed low-dose combination of two insulin sensitisers [pioglitazone (PIO) and metformin (MET), with different modes of action], and one mixed anti-androgen and anti-mineralocorticoid (spironolactone), was superior to an OC in normalising the PCOS phenotype, including ovulation rates and hepato-visceral fat.

ELIGIBILITY:
Inclusion Criteria:

1. Age range within the AYAs category (> 12.0 years and ≤ 23.9 years at study start) (96); Given that another inclusion criterium is gynaecological age (years elapsed since menarche) of 2 years or more, and that menarche before age 10.0 years is an exclusion criterium (please see exclusion criteria below), the youngest participant will be older than 12.0 years at study start (97). The upper age limit at study start is set at 23.9 years (thus, 24.9 years when the active treatment ends, see section 7. Conduct), in order to avoid early dropouts due to an increase in the prevalence of pregnancy wish beyond that age in most European countries;
2. Gynaecological age of 2 years or more;
3. Clinical androgen excess, as defined by the presence of hirsutism (modified Ferriman-Gallwey score ≥ 4) (17,98) and/or inflammatory acne (Leeds scale) unresponsive to medications (3,95,99). The scarce normative data existing in adolescents suggest that an adult level of hirsutism is reached around 2 years after menarche (100);
4. Biochemical androgen excess, as defined by increased total testosterone (≥50 ng/dL), and/or a FAI higher than 3.5 [FAI, total testosterone (nmol/L) x 100/SHBG (nmol/L)], in the follicular phase of the cycle (days 3-7) or after 2 months of amenorrhea (3,100,101); Measurements of total testosterone and/or FAI are the most recommended assessments to screen for hyperandrogenaemia (3,19,95,102). Serum testosterone attains adult levels shortly after menarche; thus, an elevation of serum testosterone concentrations and/or FAI above adult norms and assessed in reliable reference laboratories constitutes biochemical evidence of hyperandrogenism (3,19,95,100). It is accepted that this upper limit can be set at 45 ng/dL for testosterone and at 3.5 for FAI (3,95,100,101,102,103). Direct free testosterone assays, such as radiometric or enzyme-linked assays, preferably should not be used in the assessment of biochemical hyperandrogenism, as they demonstrate poor sensitivity, accuracy and precision (17);
5. Menstrual irregularity, as defined by ≤ 8 menses per year corresponding to an average inter-menstrual time of ≥45 days (3,95,100); Most adolescents establish a menstrual interval of 20-45 days within the first 2 years after menarche (3,95). Three years after menarche, the 95th percentile for cycle length is 43.6 days (104); thus, cycles longer than 45 days (<8 periods/year) at or beyond this gynaecological age are considered abnormal and are evidence of oligo-anovulation;
6. Written informed consent obtained from the patient, or assent from the patient and consent by the parents or the legally acceptable representative if she is a minor (for details, see section 7. Conduct, under informed consent).

Exclusion Criteria:

-

Ages: 12 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 364 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
On-treatment ovulation rate. | Following end of each two 12-week on-treatment periods (month 0-3 and month 9-12)
  On-treatment ovulation rate.
Post-treatment ovulation rate. | Following the end of post-treatment period (month 12-15)
  Post-treatment ovulation rate.

SECONDARY OUTCOMES:
Clinical variable: hirsutism | Every 3 months from study start to study completion (estimated 18 months)
  Presence of hirsutism as measured by the modified Ferriman & Gallwey score
Clinical variable: Acne | Every 3 months from study start to study completion (estimated 18 months)
  Presence of Acne as evaluated using the Leeds Acne Grading Scale
Clinical variable: menstrual regularity | Every 3 months from study start to study completion (estimated 18 months)
  Assessment of the menstrual regularity
Circulating androgens | Every 3 months from study start to study completion (estimated 18 months)
  Assessment by measurement of circulating androgens
Lipids | Baseline, at month 3, month 6 and month 12 whiled on treatment and 6 months after the end of treatment
  Assessment by measurement of total cholesterol, low-density lipoprotein (LDL-cholesterol), high-density lipoprotein (HDL- cholesterol), triglycerides;
Insulinaemia | Baseline and at the end of treatment (month 12) and 6 months after treatment
  Fasting and 2 hours after a 75-gr oral glucose load [oral glucose tolerance test (oGTT). Estimation of insulin resistance from fasting insulin and glucose levels using the homeostasis model assessment (HOMA);
Inflammation markers | Baseline and at the end of treatment (month 12) and 6 months after treatment
  Inflammation markers
Insulin sensitivity | Baseline and at the end of treatment (month 12) and 6 months after treatment
  Insulin sensitivity
Ultra-sensitive C-reactive protein (us-CRP); | Baseline, at month 3, month 6 and month 12 whiled on treatment and 6 months after the end of treatment
  Ultra-sensitive C-reactive protein (us-CRP);
Growth-and- differentiation factor-15 (GDF15); | Baseline, at month 3, month 6 and month 12 whiled on treatment and 6 months after the end of treatment
  Growth-and- differentiation factor-15 (GDF15);
High molecular weight adiponectin (HMW-adip), | Baseline, at month 3, month 6 and month 12 whiled on treatment and 6 months after the end of treatment
  High molecular weight adiponectin (HMW-adip),
C-X-C motif chemokine ligand 14 (CXCL14) (69,81); | Baseline, at month 3, month 6 and month 12 whiled on treatment and 6 months after the end of treatment
  C-X-C motif chemokine ligand 14 (CXCL14) (69,81);
Epigenetic variable | Baseline, at month 3, month 6 and month 12 whiled on treatment and 6 months after the end of treatment
  Circulating microRNA 451-a (miR-451a) concentrations (88);
Imaging: Cardiovascular risk | Baseline, at month 3, month 6 and month 12 whiled on treatment and 6 months after the end of treatment
  As measured by ultrasound
Imaging: Body composition | Baseline and at the end of treatment (month 12) and 6 months after treatment
  As measured by dual-energy X-ray absorptiometry (DXA)
Imaging: Abdominal fat distribution (subcutaneous and visceral) | Baseline and at the end of treatment (month 12) and 6 months after treatment
  As measured by MRI
Imaging:hepatic fat | Baseline and at the end of treatment (month 12) and 6 months after treatment
  As measured by MRI
Abdominal fat distribution | Baseline and at the end of treatment (month 12) and 6 months after treatment
  Waist circumference, Waist to hip ratio (WHR), and hepatic fat by MRI
Weight | Every 3 months from study start to study completion (estimated 18 months)
  Weight measurement
Improvement of co-morbidities | Every 3 months from study start to study completion (estimated 18 months)
  Improvement of co-morbidities
Improvement of health behaviour | Every 3 months from study start to study completion (estimated 18 months)
  Improvement of health behaviour
Improvement of health-related quality of life (HRQoL) | Baseline, at month 3, month 6 and month 12 whiled on treatment and 6 months after the end of treatment
  As reported by the patient
Safety laboratory tests | Baseline, at month 3, month 6 and month 12 whiled on treatment and 6 months after the end of treatment
  Blood count, electrolyte panel, urea, alanine transaminase (ALT), aspartate transaminase (AST), gamma-glutamyltransferase (GGT), creatinine, vitamin B12 and folic acid;
Adverse events (AEs) | Every 3 months from study start to study completion (estimated 18 months)
  As reported by the patient
Adherence | Every 3 months from study start to study completion (estimated 18 months)
  Adherence will be calculated as the ratio between the number of tablets prescribed and dispensed for the period between hospital appointments and the number of tablets returned by the patient at the following appointment;
Acceptability of the treatment | Every 3 months from study start to study completion (estimated 18 months)
  Acceptability of the tablet by the study patients
PROMs (patient-reported outcomes) | Baseline, at month 3, month 6 and month 12 whiled on treatment and 6 months after the end of treatment
  Questionnaire SF-36
PROMs (patient-reported outcomes) | Baseline, at month 3, month 6 and month 12 whiled on treatment and 6 months after the end of treatment
  Questionnaire PCOSQ
HRQoL (health-related quality of life) | Baseline, at month 3, month 6 and month 12 whiled on treatment and 6 months after the end of treatment
  Questionnaire SF-36
HRQoL (health-related quality of life) | Baseline, at month 3, month 6 and month 12 whiled on treatment and 6 months after the end of treatment
  Questionnaire PCOSQ

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Ibañez, MD, PhD, Principal Investigator — Investigator
Locations (7):
- Universitätsklinik für Innere Medizin, Graz, Austria
- Odense University Hospital (UNIODE), Odense, Denmark
- Azienda Ospedaliero Universitaria di Bologna, Bologna, Italy
- St. Olavs Hospital, Trondheim, Norway
- Spain (2):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat
  - Hospital Universitari de Girona Dr. Trueta, Girona
- İstanbul Faculty of Medicine Topkapı, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No